CLINICAL TRIAL: NCT06716333
Title: The Effects of Periodic Training on Physical and Motor Performance in Wrestlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Furkan ÇAMİÇİ, Phd, Hitit University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024/07
Record Dates: First submitted 2024-11-19; First posted 2024-12-04 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Effects of 12 Weeks of Wrestling Training
Keywords: Training; Wrestling; Motor performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intensive Training Group (Experimental)
  Interventions: Other: Experimental Group (12-Week Wrestling Training)

INTERVENTIONS:
Other: Experimental Group (12-Week Wrestling Training) — The intervention consists of a structured 12-week intensive wrestling training program designed specifically for male wrestlers aged 12-14 years. This program was conducted at athlete training centers equipped with international standard facilities, and led by professional coaches. The training included 5 sessions per week, each lasting approximately 80 minutes, with a total weekly duration of 400 minutes. Each session consisted of 20 minutes of gymnastic warm-up, 50 minutes of basic technical and strength exercises (e.g., squats, push-ups, deadlifts), and 10 minutes of stretching.

SUMMARY:
The aim of this study was to investigate the effects of 12 weeks wrestling training on the physical and motor performance parameters of wrestlers in athlete training centers. The effect of 12 weeks of intensive training was investigated in 33 wrestlers aged 12-14 years in athlete training centers in Çorum province. Paired samples t-test was used in the statistical procedures.

ELIGIBILITY:
Inclusion Criteria:

Male wrestlers aged 12-14 years. Participants enrolled in athlete training centers in Çorum province. Those who have given informed consent and whose legal guardians have also provided consent.

Participants who have no physical or medical conditions preventing them from performing intense physical activity.

Participants who are actively attending training sessions during the study period.

Exclusion Criteria:

Wrestlers with chronic illnesses or injuries that could interfere with physical training.

Participants who do not regularly attend the training program. Individuals who did not provide informed consent or whose guardians did not consent.

Ages: 12 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Male
Enrollment: 33 (Actual)
Dates: Start 2024-10-18 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Effects of Periodic Training on Physical and Motor Performance in Male Wrestlers | 12 weeks
  Measurement of body weight: A Tanita digital scale was used to measure the participants' body weight.
  Height: The heights of the participants were measured in cm. Long jump from a standing position: The measurements were taken on a flat surface behind a line and the subjects were asked to jump from the point where they were standing to the furthest point with both feet.
  20 m shuttle run test: The 20 m shuttle run test was carried out according to Leger and Lambert (1982).
  30 m sprint: The 30 m sprint values of the subjects were determined by running on the tartan track with suitable running shoes through digital photocells attached to the start and end points.
  Throwing a medicine ball: Subjects were asked to throw a 2 kg medicine ball as far as possible from a point determined.
  Sit-to-lie flexibility test 30 s number of sit-ups The maximum number of sit-ups the subjects performed in 30 s with their hands behind their back and knees bent was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Wrestling Center, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data presented in this study are available on request from the corresponding author. The data are not publicly available due to restrictions related to ongoing work for further publications